CLINICAL TRIAL: NCT04050644
Title: Comparison of Treatment With Preservative-free Dexamethasone 0.1% (Monofree Dexamethason) and Diclofenac 0.1% (Dicloabak) Eye Drops Versus Preserved Dexamethasone 0.1% (Maxidex) and Diclofenac 0.1% (Voltaren Ophtha) Eye Drops After Cataract Surgery
Acronym: GIST
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Collaborators: Laboratoires Thea (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: S60915
Record Dates: First submitted 2019-08-02; First posted 2019-08-08 (Actual); Last update posted 2024-07-01 (Actual); Status verified 2024-06

CONDITIONS: Age-related Cataract
Keywords: Preservative-free ocular drops; Preserved ocular drops

STUDY DESIGN:
Intervention Model Description: * Prospective, randomized controlled trial, investigator masked.
  * Patients requiring cataract surgery and who consent to participate will be enrolled in this study.
  * The patient can opt to participate in an sub-investigation researching a correlation between the microbiome and ocular surface inflammation post cataract surgery.
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Preservative-free dexamethasone 0.1%/diclofenac 0.1% (Experimental): One week before surgery, patients will be randomized to either receive the preservative-free dexamethasone 0.1% and diclofenac 0.1% eye drops.
  Interventions: Drug: Preservative Free drop treatment
- Preserved dexamethasone 0.1%/diclofenac 0.1% (Active Comparator): One week before surgery, patients will be randomized to either receive the preserved dexamethasone 0.1% and diclofenac 0.1% eye drops.
  Interventions: Drug: Preserved drop treatment

INTERVENTIONS:
Drug: Preservative Free drop treatment — Patients will use the preservative-free dexamethasone 0.1% 4 times a day in the first week after cataract surgery, 3 times a day in the second week, twice daily in the third week and once daily in the fourth week and diclofenac 0.1% eye drops 3 times daily for 1 day preoperatively and every 15 minutes in the hour before surgery and then 3 times a day for four weeks.
  Arms: Preservative-free dexamethasone 0.1%/diclofenac 0.1%
Drug: Preserved drop treatment — Patients will use the preserved dexamethasone 0.1% 4 times a day in the first week after cataract surgery, 3 times a day in the second week, twice daily in the third week and once daily in the fourth week and diclofenac 0.1% eye drops 3 times daily for 1 day preoperatively and every 15 minutes in the hour before surgery and then 3 times a day for four weeks.
  Arms: Preserved dexamethasone 0.1%/diclofenac 0.1%

SUMMARY:
To compare treatment with preservative-free dexamethasone 0.1% (Monofree Dexamethason) and diclofenac 0.1% (Dicloabak) eye drops versus preserved dexamethasone 0.1% (Maxidex) and diclofenac 0.1% (Voltaren Ophtha) eye drops after cataract surgery in terms of postoperative inflammation, iatrogenic dry eye disease and cystoid macular edema.

DETAILED DESCRIPTION:
Cataract surgery is a standardized procedure yielding excellent visual outcomes in most patients. According to Daien et al., the incidence of cataract surgery in 2012 in France was 11/1000 person-years. Although there are few complications related to the surgery, patients often experience ocular discomfort in the postoperative period.

Postoperative treatment usually includes topical non-steroidal anti-inflammatory drugs and topical steroids for four weeks to control anterior chamber inflammation, to relieve ocular pain after surgery and to reduce the incidence of cystoid macular edema.

Benzalkonium chloride (BAK) is the most common eye drop preservative and is associated with several ocular adverse effects, including dry eye and ocular surface inflammation. Moreover, in two clinical trials comparing the effects of BAK-containing and preservative-free eye drops, anterior chamber inflammation was reported in response to BAK after 1 month of exposure. Finally, besides the fact that intra-ocular inflammation increases the risk of macular edema, there is some evidence in the literature suggesting that BAK may also contribute to the development of macular edema.

Because of these well-established detrimental effects of preservatives, pharmaceutical industry has invested in the development of preservative-free eye drops in the past decade, which has led to preservative-free alternatives for almost all the eye medications.

The aim of this project is to investigate whether omitting preservatives from the postoperative topical treatment after cataract surgery can reduce symptoms and signs of ocular surface disease, intra-ocular inflammation and the incidence of cystoid macular edema.

Additionally ocular microbiome research is added to our study because of its known correlation with the ocular immunity. Although the ocular surface is continuously colonized by a commensal microbial community, the healthy ocular surface is not in an inflammatory state. This phenomenon suggests that there is an interplay between the ocular surface microbiome and innate immune mechanisms, which prevents inflammatory responses against commensal microbiota.

St Leger et al. used a murine model to reveal the presence of a commensal, Corynebacterium mastitidis, on the ocular surface. Corynebacterium mastitidis elicited an IL-17 response from ƔΔT-cells, facilitating recruitment of neutrophils to the ocular surface and secretion of antimicrobial peptides in the tears. These findings suggest the presence of a functional resident microbiome on the ocular surface which contribute to immune homeostasis and protects the ocular surface from pathogens.

Our expert in the area of ocular microbiome research is affiliated with the department of biochemistry and microbiology of the University of Ghent.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with age-related cataract
* Age 60 years or above

Exclusion Criteria:

* Unwilling to sign informed consent
* Pseudoexfoliation syndrome
* Functionally monocular patient
* Any use of eye drops during at least 3 months before surgery with the exception of artificial tears
* Pre-existing dry eye disease according to the criteria's of the TFOS DEXS II report
* Previous ocular surgery, laser treatment or uveitis, with the exception of retinal laser treatment (more than 6 months ago) and iridotomy (more than 6 months ago)
* Active conjunctivitis
* Wearing of contact lens
* Presence of any macular diseases possibly impacting visual acuity
* Presence of any ocular diseases leading to difficulty to have a correct eye examination
* Known or suspected allergy to any of the ingredients on the study medications
* Presence of uncontrolled systemic disease

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2018-10-30 (Actual); Primary Completion 2024-06 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
The superiority of treatment arm without conservative (WC) on treatment arm with conservative (C) on the aqueous flare value in the operated eye, measured with a laser flare meter, at week 4 after cataract surgery. | 4 weeks
  The Laser Flaremeter can measure the protein density in the anterior chamber by counting the photons. Flare Value is expressed in photoncount/ms. 1-9 photoncounts/ms is a normal value. Photoncount/ms from 10-500 is abnormal and indicates an inflamed eye.

SECONDARY OUTCOMES:
Tear Osmolarity | 4 weeks
  The difference in Tear Osmolarity between the two treatment arms. Tear Osmolarity value will be measured with TearLab.
Conjunctival Hyperemia | 4 weeks
  The difference in Conjunctival Hyperemia between the two treatment arms. The scale that will be used is the Cornea and Contact Lens Research Unit (CCLRU) scale. Minimum score is 1, maximum score is 4.
Corneal Fluorescein Staining | 4 weeks
  The difference in Corneal Fluorescein Staining between the two treatment arms. The grading scale that will be used is the Oxford grading scale. Minimum score is grade 0, maximum score is grade 5.
Tear-film break up time | 4 weeks
  The difference in Tear-film break up time between the two treatment arms. The Tear-film break up time will be expressed in seconds.
Corneal Sensitivity | 4 weeks
  The difference in Corneal Sensitivity between the two treatment arms. Corneal Sensitivity value will be measured with the Cochet-Bonnet Aesthesiometer, expressed in mm.
Central macular thickness | 4 weeks
  The difference in Central Macular Thickness between the two treatment arms. Central Macular Thickness will be measured with OCT Cirrus, expressed in µm.
DEQ-5 score | 4 weeks
  The difference in Five-item Dry Eye Questionnaire (DEQ-5) score between the two treatment arms. Minimum total score is 0, maximum total score is 22.
Inflammatory cytokine activities in tears | 4 weeks
  The difference in Inflammatory cytokine activities in tears between the two treatment arms. The cytokines that will be measured are IL-1Bèta, TNF-Alpha, IL-6, IL-8, IL-17, INF γ, macrophage migration inhibitory factor,...
Amount of tears | 4 weeks
  The difference in Amount of Tears between the two treatment arms. The Amount of Tears will be measured with Schirmer tear test strips. The strips will be placed in the lower eyelid pouch for 5 minutes, value is expressed in mm.

CONTACTS AND LOCATIONS:
Overall Officials: Heleen Delbeke, MD, Principal Investigator — Universitaire Ziekenhuizen KU Leuven
Locations (2):
- Belgium (2):
  - Universitaire Ziekenhuizen Leuven, Leuven, Vlaams-Brabant
  - AZ Delta, Roeselare, West-Vlaanderen